CLINICAL TRIAL: NCT05733039
Title: Association of Expectations and Pain Relief After Diagnostic Nerve Blocks (EXPECT) - a Prospective Cohort Study
Brief Title: Association of Expectations and Pain Relief After Diagnostic Nerve Blocks
Acronym: EXPECT
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Michael Harnik, Dr. med., senior physician, Insel Gruppe AG, University Hospital Bern
Other Study IDs: EXPECT 2021-00459
Record Dates: First submitted 2022-07-14; First posted 2023-02-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pain; Expectations
Keywords: Pain; Expectations; Local anaesthetic; Pain treatment
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Expectations are a major driver of changes in health-related outcomes and are related to reduced pain after medical treatment. However, no studies have specifically addressed the role of expectations in connection with the success of interventional pain techniques and the specific effect of expectations on diagnostic and therapeutic procedures in this field. Further, there are no studies on prolonged pain reduction after diagnostic nerve blocks. This prospective cohort study will investigate patients' outcome-related expectations measured by validated questionnaires (i.a. the Expectation for Treatment Scale) before standardized diagnostic nerve blocks (i.e. lumbar medial branch and greater occipital nerve blocks) and their association with immediate pain reduction, calculated using a numeric rating scale (NRS) before and after the block. Secondary outcomes are specificity of pain relief duration in relation to the local anesthetic, changes in pain-related interference, quality of life and function, as well as patients' global impression of change after one week in order to assess possible therapeutic effects of the nerve blocks themselves. The sample size of 110 patients is based on a power of 80% and a significance level of 0.05. Additional endpoints will be evaluated using mixed-effects linear regression, non-linear relationships between expectation and endpoints will be modelled using fractional polynomials. This research will quantify the effect of patients' expectations on pain reduction after nerve blocks, extend our knowledge which patients are likely to respond to interventional pain treatments and under which circumstances nerve blocks may exhibit therapeutic effects.

DETAILED DESCRIPTION:
Expectations are a major driver of change in health-related outcomes and are related to reduced pain after medical treatment. However, studies on expectations and their relation to pain relief after nerve blocks are largely lacking and there is a paucity of high-quality research in this area. These blocks are frequently used in interventional pain therapy to confirm a particular diagnosis (diagnostic blocks), and to predict if a patient could profit from a particular therapy (prognostic blocks). To current knowledge, there are no studies that specifically assess the association of expectation and response to pain relief after nerve blocks. A further aspect is longer lasting pain relief (i.e. sometimes for days or even weeks) that is sometimes observed in clinical practice after diagnostic nerve blocks and often attributed to a placebo effect. This may lead clinicians to perform block "series" in a therapeutic attempt. Such efforts can be controversial, since the duration of action of local anesthetics is limited to a few hours only - e.g. typically to 2-4 hours in the case of lidocaine, a short acting amino amide and one of the most widely used substances.

There are no investigations on prolonged pain relief after nerve blocks and despite decades of their use in clinical practice, there is hardly any research available.

Hypothesis and primary objective The investigators' goal is to evaluate the association of patients' outcome-related expectations with the short-term success of diagnostic blocks and to assess whether expectations contribute to longer-lasting therapeutic effects. Therefore, they will conduct a prospective cohort study of patients receiving diagnostic nerve blocks in our tertiary pain clinic. According to current recommendations on clinical outcome assessment, pain intensity, physical functioning, emotional functioning and ratings of improvements are all collected. We hypothesize that expectations play a major role in the extent of pain relief in % as well as its duration after the application of local anesthetics, i.e. in this case longer than 2-4 hours for lidocaine.

They will also analyze other potentially influential factors such as depressive symptoms, anxiety and catastrophizing - these are secondary objectives. Thus, they aim to quantify the effect of expectations, assess the therapeutic potential of nerve blocks, improve the accuracy of pretests and exclude patients from clinical pathways who are unlikely to profit from them.

ELIGIBILITY:
Inclusion Criteria:

* referral to our pain clinic
* interventions: Lumbar medial branch block or greater occipital nerve block, both with lidocaine 2%

Exclusion Criteria:

* Psychiatric co-morbidities other than depression
* Inability to express pain scores on a numeric rating scale
* Refusal of informed consent
* Insufficient knowledge of German, French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All referred pain patients (acute and chronic), scheduled for a first diagnostic nerve block.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | 30 minutes
  Change in pain intensity directly after the diagnostic nerve block, calculated on an 11-point numeric rating scale (NRS 0-10, 0=no pain; 10=unbearable pain) before and 30 minutes after the nerve block.

SECONDARY OUTCOMES:
Change in pain intensity (longterm) | 1 week
  Change in pain intensity on the same day and during one week after diagnostic block, calculated on an 11-point numeric rating scale (NRS 0-10, 0=no pain; 10=unbearable pain).
Specificity of local anesthetic | 1 day
  Specificity of local anesthetic within one day after diagnostic block (duration of pain relief corresponds to substance: yes/no)
Pain-related disability after 1 week | 1 week
  Pain-related disability using the Brief Pain Inventory: Pain severities for worst, least, average and actual pain are calculated on an 11-point numeric rating scale (NRS 0-10, 0=no pain; 10=unbearable pain). The 7 interference items (sleep disturbance, general activity, mood, work, relations with others, walking, and enjoyment of life) are assessed on a 0-10 scale, with 0 being "did not interfere" and 10 being "interfered completely.
Patient Global Impression of Change (PGIC) after 1 week | 1 week
  Patient Global Impression of Change (PGIC) one week after diagnostic block with the items "pain intensity", "quality of life" and "ability to function", measured on a 7-point scale (1="very much better", 7="very much worse")

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harnik, Dr. med., Principal Investigator — Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospital, Bern, Canton of Bern, Switzerland